CLINICAL TRIAL: NCT07122674
Title: Prospective Clinical Study of 18F-Pentixafor PET Imaging in Hematologic Malignancies
Brief Title: 18F-Pentixafor PET in Hematologic Malignancies
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: FAHZU-CXCR4-Hemic
Record Dates: First submitted 2025-08-07; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-05

CONDITIONS: Hematological Malignancies
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 18F-Pentixafor PET/CT in Hematologic Malignancies: Each patient receive a single intravenous injection of 18F-Pentixafor 55 MBq/kg and undergo PET/CT or PET/MR scan after 60 min post-injection.
  Interventions: Drug: 18F-Pentixafor

INTERVENTIONS:
Drug: 18F-Pentixafor — Patients with hematological malignancies receive 55 MBq/kg of 18F-Pentixafor intravenously followed by PET/CT or PET/MR after 60min of injection.

SUMMARY:
The aim of this study is to evaluate the efficacy of 18F-Pentixafor PET imaging in the diagnosis, staging and response evaluation of hematological malignancies.

DETAILED DESCRIPTION:
18F-FDG PET imaging based on the principle of glucose metabolism imaging is currently dominant in the staging and efficacy evaluation of lymphoma, but it is not suitable for a wider range of hematological tumors. Chemokine receptor 4 (CXCR-4) is a G protein-coupled receptor, which is overexpressed in a variety of hematological malignancies (MM, leukemia, lymphoma, etc.). It promotes tumor growth, invasion, metastasis, drug resistance, immune escape, and is associated with poor prognosis of tumors. 18Fluorine18 (18F)-NOTA-Pentixafor (18f-pentixafor) is a novel specific molecular probe targeting CXCR-4. Compared with 68Ga-Pentixafor, 18f-pentixafor has a longer half-life. More patients can be used in one synthesis, and the image quality is better and the spatial resolution is higher. Patients can undergo PET at 1 h after injection without special preparation. The aim of this study is to evaluate the performance of 18F-Pentixafor PET imaging in the diagnosis, staging, and response evaluation of hematological malignancies. Patients with suspected or histologically confirmed hematological malignancies will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18-80 years old, both sexes, with behavioral capacity;
2. patients with suspected or confirmed hematological malignancies;
3. 18F-FDG PET or other imaging examinations should be performed according to the treatment plan;
4. For suspected patients, biopsy or needle biopsy is expected to obtain pathological results;
5. Can provide informed consent, can understand and comply with the requirements of the study.

Exclusion Criteria:

1. pregnant and lactating women;
2. patients with fear or radiophobia, or with mental disorder or primary affective disorder;
3. received ionizing radiation outside the scope of this study for clinical medical or scientific research purposes within the past year, resulting in an annual radiation exposure dose exceeding 50 mSv;
4. received investigational drugs or devices of uncertain efficacy or safety within 1 month;
5. Any condition that the chairpersons of the study consider that any link related to the study may cause harm or have potential harm.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with suspected or confirmed Hematologic Malignancies
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Diagnostic efficacy | through study completion, an average of 1.5 year
  Sensitivity, specificity, positive and negative predictive value of 18F-Pentixafor PET/CT and PET/MR Imaging in hematological malignancies.

SECONDARY OUTCOMES:
18F-Pentixafor PET performence compared with 18F-FDG | up to 24 months
  Differences in sensitivity and specificity: McNemar test Differences in AUC values: DeLong test Detection rate of lesions: chi-square test. SUVmax/TBR difference: Paired t-test (normal distribution) or Wilcoxon signed-rank test (non-normal) Correlation analysis: Spearman's rank correlation was used to assess the correlation of uptake between the two imaging methods.
  Subgroup analysis: Chi-square test or Logistic regression was used to analyze heterogeneity in diagnostic power stratified by disease type and stage.
Deauville Score | through study completion, 3-4 years
  1. Score consistency analysis Agreement with 18F-FDG: Calculated agreement between the two imaging scores for the same patient (percentage agreement & Cohen's Kappa).
  2. correlation between scores and clinical outcomes Prediction of treatment response: use the International Working Group criteria (Lugano classification) as the gold standard (complete response CR, partial response PR, etc.) The association between 18F-Pentixafor scores (e.g., DS≤3 vs. DS≥4 after treatment) and treatment response (chi-square test) was calculated.
     Prognostic Value: Analyze the association of 18F-Pentixafor score (e.g., baseline DS≥4) with progression-free survival (PFS) or overall survival (OS) (Cox proportional-hazards model). The prognostic efficacy of 18F-Pentixafor and 18F-FDG scoring was compared (area under the ROC curve, AUC).
  3. score critical value optimization:If the physiological profiles of 18F-Pentixafor and 18F-FDG differ significantly (e.g., higher hepatic uptake), explore adjusted cutoffs

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China